CLINICAL TRIAL: NCT01824862
Title: Reduction of Foveal Sensitivity in Eyes With Diabetic Macular Oedema, With and Without Centre Involvement
Brief Title: Reduction of Foveal Sensitivity in Eyes With Diabetic Macular Edema
Status: Completed | Type: Observational
Sponsor: Hospital Juarez de Mexico (Other Government)
Responsible Party: Principal Investigator, Virgilio Lima Gomez, PhD, Hospital Juarez de Mexico
Other Study IDs: HJM2021/11-B
Record Dates: First submitted 2013-03-26; First posted 2013-04-05 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Diabetic Retinopathy; Clinically Significant Macular Edema
Keywords: clinically significant macular edema; foveal thickness; foveal sensitivity; perimetry; diabetic retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- eyes without diabetic retinopathy: eyes of patients with diabetes mellitus type 2 that does not have retinopathy
- CSME without centre involvement: eyes with CSME without thickening in the 500 µm adjacent to the centre of the macula
- CSME with centre involvement: eyes with CSME with thickening in the 500 µm adjacent to the centre of the macula

SUMMARY:
Clinically significant macular edema (CSME) is a thickening of the macula associated with the risk of visual loss, which increases its centre is involved. Functional evaluation of the macula relies on best corrected visual acuity; however, neural dysfunction in diabetic eyes appears before retinal thickening and visual loss. Retinal sensitivity decreases in eyes with CSME, but it is unknown whether it differs between eyes with and without centre thickening.

Aim: To compare the reduction of foveal sensitivity in eyes with CSME, with and without centre thickening.

DETAILED DESCRIPTION:
A non-experimental, comparative, prospective, cross-sectional study was conducted. Target population were type 2 diabetics, from Mexico City and its metropolitan area, and available population were type 2 diabetics who attended an Ophthalmology service from a general hospital in Mexico City, from September 2011 to May 2012.

Type 2 diabetic patients aged 30-85 years, from any gender, with central fixation, whose ocular media allowed obtaining an adequate quality Optical Coherence Tomography, who had CSME with focal angiographic pattern were included. Eyes with optic nerve or visual pathways diseases or any other ocular disease that decreased Best corrected visual acuity, were excluded. Diabetic patients without retinopathy who fulfilled the remaining selection criteria were evaluated as the reference group.

Sixty degrees colour fundus photographs were obtained in all the patients using a Visucam lite ocular fundus camera; in group 1 it was verified that no signs of diabetic retinopathy existed in the photographs; CSMO was diagnosed by biomicroscopy under mydryasis, according to the ETDRS criteria.

Retinal thickness was measured using Stratus optical coherence tomography (OCT), version 4.0.1 (Zeiss). The 6 mm fast macular map strategy was used, according to the following standardised operating procedure: mydriasis ≥6mm, inclusion of the spherical equivalent and anteroposterior axis, and optimisation of z axis and of polarisation; the photograph was taken with flash between 9:00 and 11:00, using an acquisition strategy for dark irises. The maps were obtained by the same investigator, independent from the one who evaluated the patients clinically; any deviation of the OCT line regarding the actual retina boundary was considered as a measurement error.

A 10° macular perimetry was obtained in all the patients, using a Humphrey field analyser model 750i (software version 4.1); the sixteen points evaluated were arbitrarily labelled. Retinal thickness within 3 mm from the centre of the fovea was measured in 9 fields, according to the fast macular map.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients
* aged 30-85 years
* from any gender
* with central fixation
* ocular media allowed obtaining an adequate quality Optical coherence tomography
* CSME with focal angiographic pattern

Exclusion Criteria:

* optic nerve or visual pathways diseases or any other ocular disease that decreased Best corrected visual acuity

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: target population were type 2 diabetics, from Mexico City and its metropolitan area, and available population were type 2 diabetics who attended an Ophthalmology service from a general hospital in Mexico City, from September 2011 to May 2012
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
foveal sensitivity | 1 day
  the ability of the fovea to perceive a light stimulus in 16 central points, which is measured in dB with a 10 degree central macular perimetry

SECONDARY OUTCOMES:
Retinal thickness | 1 day
  measured in µm, according to the automatic value generated by the fast macular map of the optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: VIRGILIO LIMA GOMEZ, PhD, Study Chair — Hospital Juarez de Mexico; Dulce M Razo Blanco Hernandez, MSc, Principal Investigator — Hospital Juárez de México
Locations (1):
- Virgilio Lima Gomez, Mexico City, Mexico City, Mexico